CLINICAL TRIAL: NCT03591744
Title: Phase 1 Study of Daratumumab When Given in Combination With Bortezomib, Dexamethasone, Doxil, and Lenalidomide in Patients With Plasma Cell Leukemia
Brief Title: Daratumumab, Bortezomib, Dexamethasone, Pegylated Liposomal Doxorubicin Hydrochloride, and Lenalidomide in Treating Participants With Plasma Cell Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Budgetary constraints
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18162; NCI-2018-01405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18162 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Plasma Cell Leukemia
MeSH Terms: conditions — Leukemia, Plasma Cell | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (daratumumab, bortezomib, chemotherapy) (Experimental): Participants receive daratumumab IV on days 1, 8, 15, and 22, dexamethasone IV/PO on days 1, 2, 8, 9, 15, 16, 22, and 23, pegylated liposomal doxorubicin hydrochloride IV on day 8, lenalidomide PO daily on days 1-14, and bortezomib SC on days 1, 4, 8, and 11 of courses 1 and 2. Participants then receive daratumumab IV on days 1, and 15, dexamethasone IV/PO on days 1, 2, 8, 9, 15, 16, 22, and 23, pegylated liposomal doxorubicin hydrochloride IV on day 8, lenalidomide PO daily on days 1-14, and bortezomib SC on days 1, 4, 8, and 11 of courses 3 and 4. Courses repeat every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Participants may receive up to 8 courses at the discretion of treating physician.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Lenalidomide; Drug: Pegylated Liposomal Doxorubicin Hydrochloride

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Dexamethasone — Given IV and PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposome; doxorubicin hydrochloride liposome; Duomeisu; Evacet; LipoDox; Liposomal Adriamycin; liposomal doxorubicin hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99

SUMMARY:
This phase I trial studies side effects of daratumumab, bortezomib, dexamethasone, pegylated liposomal doxorubicin hydrochloride, and lenalidomide in treating participants with plasma cell leukemia. Monoclonal antibodies, such as daratumumab, may interfere with the ability of cancer cells to grow and spread. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as, dexamethasone, pegylated liposomal doxorubicin hydrochloride, and lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving daratumumab, bortezomib, dexamethasone, pegylated liposomal doxorubicin hydrochloride, and lenalidomide in treating participants with plasma cell leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose(s) (MTD)/recommended phase 2 dose(s) (RP2D) of, bortezomib and pegylated liposomal doxorubicin hydrochloride (doxil) when given in combination with fixed dose daratumumab, lenalidomide, and dexamethasone.

SECONDARY OBJECTIVES:

I. To assess the tolerability and safety of the planned regimen, by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

II. To estimate and assess overall response rate, response duration, and survival probabilities (overall and progression-free).

EXPLORATORY OBJECTIVES:

I. Quantify CD38+ cells from the peripheral blood mononuclear cells (PBMC) fraction, including T, natural killer (NK), and monocytic subsets.

II. Assess possible changes in CD38 expression, as well as the co-receptor marker CD31, overall and by response status (responder/non-responder).

III. Assess cytokine levels in peripheral blood plasma. IV. Quantify CD38+ cells from the bone marrow CD-138 negative fractions and acellular fractions, including T, NK, and monocytic subsets.

V. Assess possible changes in CD38 expression, as well as the co-receptor marker CD31, overall and by response status (responder/non-responder).

VI. Assess cytokine levels in the bone marrow acellular fraction. VII. Investigate CD38 cellular localization in plasma cells and extracellular vesicles from blood plasma.

VIII. Assess messenger ribonucleic acid (mRNA) expression in the peripheral blood mononuclear cell (PBMC), the bone marrow CD138-negative fraction, the T cell fraction, and plasma cells.

IX. Investigate epigenetic changes in CD38 mRNA expression.

OUTLINE:

Participants receive daratumumab intravenously (IV) on days 1, 8, 15, and 22, dexamethasone IV/orally (PO) on days 1, 2, 8, 9, 15, 16, 22, and 23, pegylated liposomal doxorubicin hydrochloride IV on day 8, lenalidomide PO daily on days 1-14, and bortezomib subcutaneously (SC) on days 1, 4, 8, and 11 of courses 1 and 2. Participants then receive daratumumab IV on days 1, and 15, dexamethasone IV/PO on days 1, 2, 8, 9, 15, 16, 22, and 23, pegylated liposomal doxorubicin hydrochloride IV on day 8, lenalidomide PO daily on days 1-14, and bortezomib SC on days 1, 4, 8, and 11 of courses 3 and 4. Courses repeat every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Participants may receive up to 8 courses at the discretion of treating physician.

After completion of study treatment, participants are followed up at 30 days and then every 3 months for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative. Assent, when appropriate, will be obtained per institutional guidelines.
* Willingness to provide bone marrow and peripheral blood samples for research purposes. If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategies (REMS) program and be willing to comply with its requirements.
* Karnofsky performance status (KPS) > 60.
* Plasma cell leukemia; either newly diagnosed or relapsed: defined as the presence of > 2 x 10^9/L peripheral blood plasma cells or plasmacytosis accounting for > 20% of the differential white cell count.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Absolute neutrophil count (ANC) >= 500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary ot disease involvement.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Total bilirubin =< 2.0 x ULN (unless has Gilbert's disease).
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Aspartate aminotransferase (AST) =< 3.0 x ULN.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Alanine aminotransferase (ALT) =< 3.0 x ULN.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Left ventricular ejection fraction (LVEF) > 45%
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Hemoglobin >= 8.0 g/dL

  * Note: Transfusion support is allowed.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Seronegative for human immunodeficiency virus (HIV) antigen-antibody (Ag/Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (RPR).

  * If positive, hepatitis C RNA quantitation must be performed.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Meets other institutional and federal requirements for infectious disease titer requirements.

  * Note: Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy.
* Within 14 days prior to day 1 of protocol therapy unless otherwise stated: Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).
* Women of childbearing potential must follow pregnancy testing requirements as outline in REMS program material.

Exclusion Criteria:

* Progression or intolerance to daratumumab, bortezomib, or lenalidomide.
* Prior stem cell transplant.
* Participant is receiving concurrent chemotherapy or biologic or hormonal therapy for cancer treatment.

  * Note: Concurrent use of hormones for noncancer-related conditions (e.g., insulin for diabetes) is acceptable.
* Vaccination with live attenuated vaccines within 4 weeks of first study agent administration.
* Participant is currently using or has used immunosuppressive medication within 14 days prior to the first study dose of study treatment. The following are exceptions:

  * Intranasal, topical, inhaled, or local steroid injections (e.g., intra-articular injection)
  * Chronic systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., infusion-related reactions, computed tomography [CT] scan premedication).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Has known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal.
* Has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification.
* Clinically significant uncontrolled illness.
* Active infection requiring intravenous antibiotics or antifungals within 14 days prior to start of study treatment.
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection.
* Grade >= 3 peripheral neuropathy, or grade >= 2 with pain on clinical examination during the screening period.
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months. Note: Prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant.
* Other active malignancy. Exceptions: Non-melanoma skin cancer, ductal breast carcinoma in situ (DCIS) or carcinoma-in-situ of the cervix. Note: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer. Prior malignancy treated with curative intent is not an exclusion.
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-25 (Estimated); Primary Completion 2019-10-25 (Estimated); Study Completion 2019-10-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 30 days
  Observed toxicities will be tabulated using frequencies and percentages based on the CTCAE v5.0.

SECONDARY OUTCOMES:
Overall response rate described by the International Myeloma Working Group (IMWG) | Up to 18 months
  Response rates will also be evaluated based on number and type of prior therapy(ies); the exact binomial confidence interval (CI) will be calculated for these estimates.
Duration of response | Up to 18 months
  The overall response rate (ORR) will be estimated by the number of participants who achieve a confirmed response (stringent complete response [sCR]/complete response [CR]/very good partial response [VGPR] or partial response [PR]) divided by the total number of response evaluable participants. Response rates will also be evaluated based on number and type of prior therapy(ies); the exact binomial CI will be calculated for these estimates.
Overall survival rate | From date of first dose of study drug to date of death from any cause, assessed up to 18 months
  Will be estimated using the product-limit method of Kaplan and Meier; 95% confidence intervals will be calculated using Greenwood's formula.
Progression-free survival rate | From date of first dose of study drug to date of first documented disease relapse, progression or death from any cause, whichever occurs first, up to 18 months
  Will be estimated using the product-limit method of Kaplan and Meier; 95% confidence intervals will be calculated using Greenwood's formula.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Krishnan, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee